CLINICAL TRIAL: NCT02787551
Title: A 26-Week Randomized, Open-label, Active Controlled, Parallel-group, Study Assessing the Efficacy and Safety of the Insulin Glargine/Lixisenatide Fixed Ratio Combination in Adults With Type 2 Diabetes Inadequately Controlled on GLP-1 Receptor Agonist and Metformin (Alone or With Pioglitazone and/or SGLT2 Inhibitors), Followed by a Fixed Ratio Combination Single-arm 26-Week Extension Period
Brief Title: Efficacy and Safety of the Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) Versus GLP-1 Receptor Agonist in Patients With Type 2 Diabetes, With a FRC Extension Period
Acronym: LixiLan-G
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC13794; 2014-004850-32; U1111-1168-4639 (Other: UTN)
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Results first posted 2019-06-12 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; lixisenatide; Liraglutide; Exenatide; rGLP-1 protein; dulaglutide; Metformin; Pioglitazone; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) (Experimental): Core period: FRC injected subcutaneously once daily (QD) for 26 weeks on top of oral anti-diabetic drug (OAD) therapy. Dose individually adjusted.
  Single arm extension period: Participants who completed core treatment period and met eligibility criteria entered in extension treatment period and received same treatment (FRC injected subcutaneously QD on top of OAD therapy) for 26 weeks (up to Week 52). Dose individually adjusted.
  Interventions: Drug: Insulin glargine/lixisenatide fixed ratio combination; Drug: Background therapy: Oral Anti-diabetic Drug (Metformin, Pioglitazone, SGLT2 inhibitor)
- GLP-1 Receptor Agonist (Active Comparator): Core period: GLP-1 RA receptor agonist (liraglutide QD, exenatide twice daily [BID], exenatide extended-release QW, albiglutide QW, or dulaglutide QW) injected subcutaneously for 26 weeks on top of OAD therapy. GLP-1 RAs were administered as per local labeling at the same dose schedule as prior to randomization.
  Interventions: Drug: liraglutide; Drug: exenatide; Drug: exenatide extended-release; Drug: albiglutide; Drug: dulaglutide; Drug: Background therapy: Oral Anti-diabetic Drug (Metformin, Pioglitazone, SGLT2 inhibitor)

INTERVENTIONS:
Drug: Insulin glargine/lixisenatide fixed ratio combination — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Other Names: HOE901/AVE0010; Soliqua
  Arms: Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC)
Drug: liraglutide — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Other Names: Victoza
  Arms: GLP-1 Receptor Agonist
Drug: exenatide — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Other Names: Byetta
  Arms: GLP-1 Receptor Agonist
Drug: exenatide extended-release — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Other Names: Bydureon
  Arms: GLP-1 Receptor Agonist
Drug: albiglutide — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Other Names: Tanzeum
  Arms: GLP-1 Receptor Agonist
Drug: dulaglutide — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Other Names: Trulicity
  Arms: GLP-1 Receptor Agonist
Drug: Background therapy: Oral Anti-diabetic Drug (Metformin, Pioglitazone, SGLT2 inhibitor) — Pharmaceutical form: tablet Route of administration: oral If previously taken, doses to remain stable through the study.

SUMMARY:
Primary Objective:

To demonstrate the superiority of the insulin glargine/lixisenatide fixed ratio combination (FRC) versus GLP-1 receptor agonist (GLP-1 RA) in hemoglobin A1c (HbA1c) change.

Secondary Objectives:

To compare the overall efficacy and safety of the insulin glargine/lixisenatide FRC to GLP-1 RA on top of metformin (with or without pioglitazone, with or without sodium-glucose co-transporter 2 [SGLT2] inhibitor) in participants with type 2 diabetes.

To evaluate safety, efficacy and other endpoints of FRC up to the end of the extension period.

DETAILED DESCRIPTION:
The maximum duration for GLP1-RA participants was approximately 29 weeks: up to 2 week screening period, a 26 week treatment period (either randomized or uncontrolled), and a 3 or 9 day post-treatment safety follow-up period.

Maximum duration for FRC participants was approximately 55 weeks: up to 2-week screening period, a 26-week randomized treatment period, a 26-week extension period and a 3-day post-treatment safety follow-up period.

All primary and secondary efficacy, safety and other outcome measures were assessed at the end of the extension period.

ELIGIBILITY:
Inclusion criteria :

* Participants with type 2 diabetes mellitus diagnosed at least 1 year prior to screening visit.
* Participants who were treated with one of the following GLP-1 receptor agonists for at least 4 months prior to screening visit 1 (V1), and with stable dose for at least 3 months prior to screening visit (V1):
* Liraglutide (Victoza®) 1.8 milligram (mg) QD or 1.2 mg QD, if the 1.8 mg QD dose was not well tolerated according to the Investigator's judgment or
* Exenatide (Byetta®) 10 microgram (µg) BID or of 5 µg BID, if 10 µg BID dose was not well tolerated according to the Investigator's judgment

in combination with metformin (daily dose greater than equal to [>=] 1500 mg/day or maximum tolerated dose [MTD]), with or without pioglitazone, with or without SGLT2 inhibitor, all at stable dose for at least 3 months prior to screening.

or

Participants who were treated with stable dose of one of the following GLP-1 receptor agonists for at least 6 months prior to screening visit (V1):

* Exenatide extended-release (Bydureon®) 2 mg once weekly (QW), if well tolerated according to Investigator's judgment,
* Albiglutide (Tanzeum®) 50 mg QW or 30 mg QW, if 50 mg QW was not well tolerated according to Investigator's judgment,
* Dulaglutide (Trulicity®) 1.5 mg QW or 0.75 mg QW, if 1.5 mg QW was not well tolerated according to Investigator's judgment

in combination with metformin (daily dose ≥1500 mg/day or MTD), with or without pioglitazone, with or without SGLT2 inhibitor, all at stable dose for at least 3 months prior to screening;

-Signed written informed consent.

Exclusion criteria:

* At screening visit, age <18.
* Screening HbA1c <7% and >9%.
* Pregnancy or lactation, women of childbearing potential with no effective contraceptive method.
* Any use of antidiabetic drugs within 3 months prior to the screening visit other than those described in the inclusion criteria.
* Previous treatment with insulin in the year prior to screening visit (note: short-term treatment with insulin [<=10 days] due to intercurrent illness including gestational diabetes was allowed at the discretion of the study physician).
* Laboratory findings at the time of screening, including:
* Fasting plasma glucose (FPG) >250 mg/dL (13.9 millimoles per litre [mmol/L]),
* Amylase and/or lipase >3 times the upper limit of the normal laboratory range (ULN),
* Alanine transaminase or aspartate transaminase >3 ULN,
* Calcitonin >=20 pg/mL (5.9 pmol/L),
* Positive pregnancy test.
* Participant who had renal function impairment with estimated glomerular filtration rate <30mL/min/1.73m^2 (using the Modification of Diet in Renal Disease formula) or end-stage renal disease.
* Contraindication to use of insulin glargine, or lixisenatide or GLP-1 receptor agonist (Victoza®, Byetta®, Bydureon®, Tanzeum® or Trulicity®) according to local labeling.
* Any contraindication to metformin or pioglitazone or SGLT2 inhibitor use, according to local labeling.
* History of hypersensitivity to insulin glargine, or to any of the excipients.
* History of allergic reaction to any GLP-1 receptor agonist or to meta-cresol.
* Personal or immediate family history of medullary thyroid cancer (MTC) or genetic condition that predisposes to MTC (eg, multiple endocrine neoplasia type 2 syndromes).
* History of pancreatitis (unless pancreatitis was related to gallstones and cholecystectomy was already performed), chronic pancreatitis, pancreatitis during a previous treatment with incretin therapies, pancreatectomy.
* Body mass index <=20 or >40 kg/m^2.

Exclusion criteria for the extension period:

* Participants in the FRC arm with a rescue therapy and HbA1c >8% at week 22.
* Participants in the FRC arm who discontinued prematurely from FRC treatment before week 26.
* Participants in the GLP-1 RA treatment arm after randomization.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (124):
- United States (74):
  - Investigational Site Number 8400064, Birmingham, Alabama
  - Investigational Site Number 8400073, Fountain Hills, Arizona
  - Investigational Site Number 8400047, Phoenix, Arizona
  - Investigational Site Number 8400103, Bakersfield, California
  - Investigational Site Number 8400137, Fresno, California
  - Investigational Site Number 8400043, Huntington Park, California
  - Investigational Site Number 8400124, Lamont, California
  - Investigational Site Number 8400027, Lancaster, California
  - Investigational Site Number 8400098, Los Angeles, California
  - Investigational Site Number 8400013, Los Angeles, California
  - Investigational Site Number 8400042, Mission Hills, California
  - Investigational Site Number 8400006, Northridge, California
  - Investigational Site Number 8400021, Orange, California
  - Investigational Site Number 8400126, Rialto, California
  - Investigational Site Number 8400094, Santa Ana, California
  - Investigational Site Number 8400009, Ventura, California
  - Investigational Site Number 8400071, Denver, Colorado
  - Investigational Site Number 8400036, Denver, Colorado
  - Investigational Site Number 8400114, Jacksonville, Florida
  - Investigational Site Number 8400133, Miami, Florida
  - Investigational Site Number 8400058, Port Charlotte, Florida
  - Investigational Site Number 8400084, Tampa, Florida
  - Investigational Site Number 8400112, West Palm Beach, Florida
  - Investigational Site Number 8400045, Lawrenceville, Georgia
  - Investigational Site Number 8400096, Snellville, Georgia
  - Investigational Site Number 8400023, Springfield, Illinois
  - Investigational Site Number 8400049, Avon, Indiana
  - Investigational Site Number 8400053, Avon, Indiana
  - Investigational Site Number 8400085, Avon, Indiana
  - Investigational Site Number 8400120, Avon, Indiana
  - Investigational Site Number 8400041, Evansville, Indiana
  - Investigational Site Number 8400038, Indianapolis, Indiana
  - Investigational Site Number 8400130, Council Bluffs, Iowa
  - Investigational Site Number 8400034, Lexington, Kentucky
  - Investigational Site Number 8400091, Lexington, Kentucky
  - Investigational Site Number 8400078, Marrero, Louisiana
  - Investigational Site Number 8400032, Metairie, Louisiana
  - Investigational Site Number 8400088, New Orleans, Louisiana
  - Investigational Site Number 8400033, Baltimore, Maryland
  - Investigational Site Number 8400051, Jefferson City, Missouri
  - Investigational Site Number 8400083, Papillion, Nebraska
  - Investigational Site Number 8400044, Henderson, Nevada
  - Investigational Site Number 8400079, Albany, New York
  - Investigational Site Number 8400061, New York, New York
  - Investigational Site Number 8400123, North Massapequa, New York
  - Investigational Site Number 8400095, Staten Island, New York
  - Investigational Site Number 8400067, West Seneca, New York
  - Investigational Site Number 8400111, Yonkers, New York
  - Investigational Site Number 8400020, Morehead City, North Carolina
  - Investigational Site Number 8400065, Wilmington, North Carolina
  - Investigational Site Number 8400018, Fargo, North Dakota
  - Investigational Site Number 8400019, Columbus, Ohio
  - Investigational Site Number 8400056, Dayton, Ohio
  - Investigational Site Number 8400125, Mentor, Ohio
  - Investigational Site Number 8400099, Oklahoma City, Oklahoma
  - Investigational Site Number 8400129, Scottdale, Pennsylvania
  - Investigational Site Number 8400076, Smithfield, Pennsylvania
  - Investigational Site Number 8400104, Warwick, Rhode Island
  - Investigational Site Number 8400090, Columbia, South Carolina
  - Investigational Site Number 8400139, Austin, Texas
  - Investigational Site Number 8400001, Dallas, Texas
  - Investigational Site Number 8400118, Edinburg, Texas
  - Investigational Site Number 8400008, Houston, Texas
  - Investigational Site Number 8400109, Houston, Texas
  - Investigational Site Number 8400063, Houston, Texas
  - Investigational Site Number 8400106, Houston, Texas
  - Investigational Site Number 8400014, North Richland Hills, Texas
  - Investigational Site Number 8400089, San Antonio, Texas
  - Investigational Site Number 8400135, Schertz, Texas
  - Investigational Site Number 8400075, Shavano Park, Texas
  - Investigational Site Number 8400107, Sugar Land, Texas
  - Investigational Site Number 8400054, Orem, Utah
  - Investigational Site Number 8400025, Salt Lake City, Utah
  - Investigational Site Number 8400092, Weber City, Virginia
- Canada (4):
  - Investigational Site Number 1240003, Burlington
  - Investigational Site Number 1240006, Corunna
  - Investigational Site Number 1240002, Red Deer
  - Investigational Site Number 1240001, Vancouver
- Estonia (4):
  - Investigational Site Number 2330002, Pärnu
  - Investigational Site Number 2330003, Tallinn
  - Investigational Site Number 2330001, Tallinn
  - Investigational Site Number 2330004, Viljandi
- Germany (2):
  - Investigational Site Number 2760001, Dresden
  - Investigational Site Number 2760003, Oldenburg in Holstein
- Israel (5):
  - Investigational Site Number 3760001, Haifa
  - Investigational Site Number 3760002, Haifa
  - Investigational Site Number 3760005, Jerusalem
  - Investigational Site Number 3760006, Jerusalem
  - Investigational Site Number 3760004, Tel Aviv
- Italy (7):
  - Investigational Site Number 3800008, Bergamo
  - Investigational Site Number 3800002, Bologna
  - Investigational Site Number 3800001, Milan
  - Investigational Site Number 3800006, Milan
  - Investigational Site Number 3800005, Napoli
  - Investigational Site Number 3800004, Roma
  - Investigational Site Number 3800003, Roma
- Romania (9):
  - Investigational Site Number 6420004, Bacau
  - Investigational Site Number 6420006, Brasov
  - Investigational Site Number 6420001, Bucharest
  - Investigational Site Number 6420008, Buzău
  - Investigational Site Number 6420003, Cluj-Napoca
  - Investigational Site Number 6420002, Oradea
  - Investigational Site Number 6420009, Târgovişte
  - Investigational Site Number 6420007, Târgu Mureş
  - Investigational Site Number 6420005, Timișoara
- Slovakia (9):
  - Investigational Site Number 7030006, Bratislava
  - Investigational Site Number 7030002, Lučenec
  - Investigational Site Number 7030009, Ľubochňa
  - Investigational Site Number 7030005, Malacky
  - Investigational Site Number 7030007, Prešov
  - Investigational Site Number 7030001, Rožňava
  - Investigational Site Number 7030008, Sabinov
  - Investigational Site Number 7030004, Trenčín
  - Investigational Site Number 7030003, Žilina
- Spain (10):
  - Investigational Site Number 7240012, Alzira
  - Investigational Site Number 7240005, Barcelona
  - Investigational Site Number 7240002, Ferrol
  - Investigational Site Number 7240008, Málaga
  - Investigational Site Number 7240011, Pozuelo de Alarcón
  - Investigational Site Number 7240003, Quart de Poblet
  - Investigational Site Number 7240006, Sabadell
  - Investigational Site Number 7240007, Seville
  - Investigational Site Number 7240009, Seville
  - Investigational Site Number 7240004, Seville

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Kuruvilla DE, Mann JI, Tepper SJ, Starling AJ, Panza G, Johnson MAL. Phase 3 randomized, double-blind, sham-controlled Trial of e-TNS for the Acute treatment of Migraine (TEAM). Sci Rep. 2022 Mar 24;12(1):5110. doi: 10.1038/s41598-022-09071-6. PMID 35332216
- [Derived] Ferrannini E, Niemoeller E, Dex T, Servera S, Mari A. Fixed-ratio combination of insulin glargine plus lixisenatide (iGlarLixi) improves ss-cell function in people with type 2 diabetes. Diabetes Obes Metab. 2022 Jun;24(6):1159-1165. doi: 10.1111/dom.14688. Epub 2022 Mar 28. PMID 35257461
- [Derived] Guja C, Giorgino F, Blonde L, Ali A, Prazny M, Meier JJ, Souhami E, Lubwama R, Ji C, Rosenstock J. Concomitant iGlarLixi and Sodium-Glucose Co-transporter-2 Inhibitor Therapy in Adults with Type 2 Diabetes: LixiLan-G Trial and Real-World Evidence Results. Diabetes Ther. 2022 Jan;13(1):205-215. doi: 10.1007/s13300-021-01180-1. Epub 2021 Dec 11. PMID 34894329
- [Derived] Blonde L, Rosenstock J, Frias J, Birkenfeld AL, Niemoeller E, Souhami E, Ji C, Del Prato S, Aroda VR. Durable Effects of iGlarLixi Up to 52 Weeks in Type 2 Diabetes: The LixiLan-G Extension Study. Diabetes Care. 2021 Mar;44(3):774-780. doi: 10.2337/dc20-2023. Epub 2021 Jan 19. PMID 33468520
- [Derived] Blonde L, Rosenstock J, Del Prato S, Henry R, Shehadeh N, Frias J, Niemoeller E, Souhami E, Ji C, Aroda VR. Switching to iGlarLixi Versus Continuing Daily or Weekly GLP-1 RA in Type 2 Diabetes Inadequately Controlled by GLP-1 RA and Oral Antihyperglycemic Therapy: The LixiLan-G Randomized Clinical Trial. Diabetes Care. 2019 Nov;42(11):2108-2116. doi: 10.2337/dc19-1357. Epub 2019 Sep 17. PMID 31530665

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 112 sites in 9 countries. A total of 840 participants were screened between 06 July 2016 and 01 November 2017, of which 326 were screen failures. Screen failures were mainly due to glycated hemoglobin (HbA1c) level lesser than (<)7% or more than (>)9% at screening visit.
Pre-assignment Details: A total of 514 participants were randomized in 1:1 (Insulin Glargine/Lixisenatide fixed ratio combination [FRC] or glucagon-like peptide-1 receptor agonist [GLP-1 RA]) ratio. Randomization was stratified by values of HbA1c at screening (<8%, >=8%) & GLP-1 RA subtype at screening (once/twice daily [QD/BID], once weekly [QW] formulations).
Groups:
- Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC): Core period: FRC injected subcutaneously QD for 26 weeks on top of oral anti-diabetic drug (OAD) therapy. Dose individually adjusted.
  Single arm extension period: participants who completed core treatment period and met eligibility criteria entered in extension treatment period and received same treatment (FRC injected subcutaneously QD on top of OAD therapy) for 26 weeks (up to Week 52). Dose individually adjusted.
- GLP-1 Receptor Agonist: Core Period: GLP-1 RA receptor agonist (liraglutide QD, exenatide BID, exenatide extended-release QW, albiglutide QW, or dulaglutide QW) injected subcutaneously for 26 weeks on top of OAD therapy. GLP-1 RAs were administered as per local labeling at the same dose schedule as prior to randomization.
Period: Core Period: 26 Weeks
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) | GLP-1 Receptor Agonist
Started | 257 | 257
Treated | 255 | 256
Completed | 230 (Out of 230 participants, 206 participants entered in single arm extension period.) | 246
Not Completed | 27 | 11
Not completed — Adverse Event | 10 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Poor compliance to protocol | 2 | 0
Not completed — Withdrawal by Subject | 9 | 9
Not completed — Randomized but not treated | 2 | 1
Not completed — Other than specified | 3 | 1
Period: Extension Period:26 Weeks(Upto 52 Weeks)
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) | GLP-1 Receptor Agonist
Started | 206 (Participants who completed core period and met eligibility criteria for extension period.) | 0
Completed | 197 | 0
Not Completed | 9 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Poor compliance to protocol | 3 | 0
Not completed — Other than specified | 5 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population.
Groups:
- Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC): FRC injected subcutaneously QD for 26 weeks on top of OAD therapy. Dose individually adjusted.
- GLP-1 Receptor Agonist: GLP-1 RA receptor agonist (liraglutide QD, exenatide BID, exenatide extended-release QW, albiglutide QW, or dulaglutide QW) injected subcutaneously for 26 weeks on top of OAD therapy. GLP-1 RAs were administered as per local labeling at the same dose schedule as prior to randomization.
- Total: Total of all reporting groups
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) | GLP-1 Receptor Agonist | Total
Number analyzed (Participants) | 257 | 257 | 514
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (9.6) | 60.0 (10.3) | 59.6 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 113 | 244
  Male | 126 | 144 | 270
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian/Oriental | 3 | 4 | 7
  Black | 12 | 7 | 19
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 241 | 244 | 485
  Unknown or Not Reported' | 0 | 2 | 2
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  <30 | 71 | 69 | 140
  >=30 | 186 | 188 | 374
Duration of diabetes [Mean (Standard Deviation); unit: years] | 11.23 (7.42) | 10.95 (6.08) | 11.09 (6.78)
Hemoglobin A1C (HbA1C) [Mean (Standard Deviation); unit: percentage of HbA1c] | 7.78 (0.62) | 7.80 (0.56) | 7.79 (0.59)
Daily dose of metformin at baseline [Mean (Standard Deviation); unit: milligrams (mg)] | 1966.93 (434.56) | 2030.74 (497.15) | 1998.83 (467.54)
Daily dose of pioglitazone at baseline [Mean (Standard Deviation); unit: mg] — Population: Here, number analyzed=number of participants with available data for specified measure.
  mg
    number analyzed (Participants) | 12 | 22 | 34
    (all) | 31.25 (10.03) | 32.73 (8.83) | 32.21 (9.14)
Daily dose of SGLT2 inhibitor at baseline [Mean (Standard Deviation); unit: mg] — Population: Here, number analyzed=number of participants with available data for specified categories.
  mg
    Canagliflozin: number analyzed (Participants) | 7 | 12 | 19
    Canagliflozin | 214.29 (106.90) | 283.33 (57.74) | 257.89 (83.77)
    Empagliflozin: number analyzed (Participants) | 6 | 9 | 15
    Empagliflozin | 15.42 (7.49) | 16.67 (8.20) | 16.17 (7.67)
    Dapagliflozin: number analyzed (Participants) | 13 | 5 | 18
    Dapagliflozin | 9.62 (3.80) | 9.00 (2.24) | 9.44 (3.38)
Duration of GLP-1 receptor agonist treatment [Mean (Standard Deviation); unit: years] | 1.89 (1.76) | 1.92 (1.85) | 1.90 (1.81)
GLP-1 receptor agonist use by type at screening [Count of Participants; unit: Participants]
  Once/twice daily formulation | 153 | 154 | 307
  Once weekly formulation | 104 | 103 | 207

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1c) to Week 26: Core Period
Description: Change in HbA1c was calculated by subtracting baseline value from Week 26 value. Adjusted least squares (LS) mean and standard error (SE) were obtained from Mixed-effect model with repeated measures (MMRM) to account for missing data using all available post baseline data during the 26 week treatment period.
Time Frame: Baseline, Week 26
Population: Modified Intent-To-Treat (mITT) population:all randomized participants who had a baseline and at least 1 post-baseline assessment of any primary/secondary outcome measures, irrespective of compliance with study protocol and procedures."Overall number of participants analyzed"=participants with baseline and at least 1 post-baseline HbA1c assessment.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Groups:
- Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC): FRC injected subcutaneously QD for 26 weeks on top of oral anti-diabetic drug (OAD) therapy. Dose individually adjusted.
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) | GLP-1 Receptor Agonist
Number analyzed (Participants) | 250 | 253
percentage of HbA1c | -1.02 (0.048) | -0.38 (0.048)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) vs GLP-1 Receptor Agonist; Analysis was performed using Mixed-effect model with repeated measures (MMRM) with treatment groups, randomization strata of Week -2 HbA1c (<8.0%, >=8.0%), GLP-1 RA subtype at screening, visits, treatment-by-visit interaction, world region as fixed effects, baseline HbA1c value-by-visit interaction as a covariate. Analysis included all scheduled measurements obtained during 26-week randomized treatment period, including those obtained after IMP discontinuation/introduction of rescue medication; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; Least square (LS) mean difference = -0.64, 95% CI 2-sided [-0.770 to -0.508], Standard Error of Mean 0.067

2. Primary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1c) to Week 52: Single Arm Extension Period
Description: Change in HbA1c was calculated by subtracting baseline value from Week 52 value.
Time Frame: Baseline, Week 52
Population: Analysis was performed on mITT population who entered the extension period. Here, "Overall number of participants analyzed" = participants with baseline and at least 1 post-baseline HbA1c assessment.
Measure: Mean (Standard Error); unit: percentage of HbA1c
Groups:
- Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC): Participants who completed core treatment period and met eligibility criteria entered in extension treatment period and received same treatment (FRC injected subcutaneously QD on top of OAD therapy) for 26 weeks (up to Week 52). Dose individually adjusted.
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC)
Number analyzed (Participants) | 202
percentage of HbA1c | -1.01 (0.063)

3. Secondary Outcome: Percentage of Participants Reaching HbA1c <7% or <=6.5% at Week 26: Core Period
Description: Participants without any available HbA1c assessment at Week 26 were considered as non-responders.
Time Frame: Week 26
Population: Analysis was performed on mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) | GLP-1 Receptor Agonist
Number analyzed (Participants) | 252 | 253
percentage of participants
  HbA1c <7% | 61.9 | 25.7
  HbA1c <=6.5% | 40.5 | 9.9
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) vs GLP-1 Receptor Agonist; HbA1c <7.0%: Insulin Glargine/Lixisenatide FRC vs GLP-1 Receptor Agonist. Analysis was performed using Cochran-Mantel-Haenszel method method stratified on randomization strata of Week -2 HbA1c (<8.0%, >=8.0%), and randomization strata of GLP-1 receptor agonist subtype at screening. Hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially per pre-specified order (only HbA1c < 7% was part of testing); Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel — Threshold for significance <=0.05; Difference in percentage = 36.05, 95% CI 2-sided [28.11 to 43.99]

4. Secondary Outcome: Percentage of Participants Reaching HbA1c <7 % or <=6.5% at Week 52: Single Arm Extension Period
Description: Participants without any available HbA1c assessment at Week 52 were considered as non-responders.
Time Frame: Week 52
Population: Analysis was performed on mITT population who entered the extension period.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC)
Number analyzed (Participants) | 206
percentage of participants
  HbA1c <7% | 64.1
  HbA1c <=6.5% | 42.7

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) to Week 26: Core Period
Description: Change in FPG was calculated by subtracting baseline value from Week 26 value. Adjusted LS means and SE were obtained from MMRM to account for missing data using all available post baseline data during the 26 week treatment period.
Time Frame: Baseline, Week 26
Population: Analysis was performed using mITT population. Here, "overall number of participants analyzed" = participants with baseline and at least one post-baseline FPG assessment.
Measure: Least Squares Mean (Standard Error); unit: millimoles per litre (mmol/L)
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) | GLP-1 Receptor Agonist
Number analyzed (Participants) | 251 | 253
millimoles per litre (mmol/L) | -2.28 (0.120) | -0.60 (0.119)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) vs GLP-1 Receptor Agonist; Analysis was performed using MMRM with treatment groups, randomization strata of Week -2 HbA1c (<8.0%, >=8.0%), randomization strata of GLP-1 RA subtype at screening, scheduled visit, treatment-by-visit interaction, and world region as fixed effects, and and baseline FPG value-by visit interaction as a covariate. Testing according to the hierarchical testing procedure (continued only if previous outcome measures were statistically significant); Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -1.67, 95% CI 2-sided [-2.001 to -1.341], Standard Error of Mean 0.168

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) to Week 52: Single Arm Extension Period
Description: Change in FPG was calculated by subtracting baseline value from Week 52 value.
Time Frame: Baseline, Week 52
Population: Analysis was performed on mITT population who entered the extension period. Here, "overall number of participants analyzed" = participants with baseline and at least one post-baseline FPG assessment.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC)
Number analyzed (Participants) | 196
mmol/L | -2.27 (0.173)

7. Secondary Outcome: Change From Baseline in the Daily Average of the 7-point Self-monitored Plasma Glucose (SMPG) to Week 26: Core Period
Description: The 7-point SMPG profile was measured at the following 7 points: pre-prandial and 2 hours postprandial for breakfast, lunch, dinner and at bedtime. Two hours postprandial (breakfast, lunch and dinner) was defined as 2 hours after the start of the meal. Adjusted LS means and SE were obtained from MMRM to account for missing data using all available post baseline data during the 26 week treatment period.
Time Frame: Baseline, Week 26
Population: Analysis was performed using mITT population. Here, "overall number of participants analyzed" = participants with baseline and at least one post-baseline 7-point SMPG assessment.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) | GLP-1 Receptor Agonist
Number analyzed (Participants) | 216 | 220
mmol/L | -1.69 (0.114) | -0.67 (0.112)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) vs GLP-1 Receptor Agonist; Analysis was performed using MMRM with treatment groups, randomization strata of Week -2 HbA1c (<8.0%, >=8.0%), randomization strata of GLP-1 RA subtype at screening, scheduled visit, treatment-by-visit interaction, and world region as fixed effects, and baseline average SMPG value-by-visit interaction as a covariate. Testing according to the hierarchical testing procedure (continued only if previous outcome measures were statistically significant); Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -1.02, 95% CI 2-sided [-1.325 to -0.708], Standard Error of Mean 0.157

8. Secondary Outcome: Change From Baseline in the Daily Average of the 7-point Self-monitored Plasma Glucose (SMPG) to Week 52: Single Arm Extension Period
Description: The 7-point SMPG profile was measured at the following 7 points: pre-prandial and 2 hours postprandial for breakfast, lunch, dinner and at bedtime. Two hours postprandial (breakfast, lunch and dinner) was defined as 2 hours after the start of the meal.
Time Frame: Baseline, Week 52
Population: Analysis was performed on mITT population who entered the extension period. Here, "overall number of participants analyzed" = participants with baseline and at least one post-baseline 7-point SMPG assessment.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC)
Number analyzed (Participants) | 142
mmol/L | -1.68 (0.176)

9. Secondary Outcome: Change From Baseline in 2-Hour Postprandial Plasma Glucose (PPG) During Standardized Meal Test to Week 26: Core Period
Description: The 2-hour PPG test measured blood glucose 2 hours after eating a liquid standardized breakfast meal. Change in PPG was calculated by subtracting baseline value from Week 26 value. Missing data was imputed using last observation carried forward (LOCF).
Time Frame: Baseline, Week 26
Population: Analysis was performed on mITT population. Here, "overall number of participants analyzed" = participants with baseline and at least one post-baseline plasma glucose assessment.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) | GLP-1 Receptor Agonist
Number analyzed (Participants) | 215 | 222
mmol/L | -3.96 (0.211) | -1.11 (0.205)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) vs GLP-1 Receptor Agonist; Analysis was performed using analysis of covariance (ANCOVA) model with treatment groups, randomization strata of Week -2 HbA1c (<8.0%, >=8.0%), randomization strata of GLP-1 RA subtype (once/twice daily formulations, once weekly formulations) at screening, and world region as fixed effects and baseline 2-hour PPG value as a covariate. Testing according to the hierarchical testing procedure (continued only if previous endpoints were statistically significant); Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -2.85, 95% CI 2-sided [-3.420 to -2.279], Standard Error of Mean 0.290

10. Secondary Outcome: Change From Baseline in 2-Hour Postprandial Plasma Glucose (PPG) During Standardized Meal Test to Week 52: Single Arm Extension Period
Description: The 2-hour PPG test measured blood glucose 2 hours after eating a liquid standardized breakfast meal. Change in PPG was calculated by subtracting baseline value from Week 52 value. Missing data was imputed using LOCF.
Time Frame: Baseline, Week 52
Population: Analysis was performed on mITT population who entered the extension period. Here, "overall number of participants analyzed" = participants with baseline and at least one post-baseline plasma glucose assessment.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC)
Number analyzed (Participants) | 192
mmol/L | -4.30 (0.284)

11. Secondary Outcome: Change From Baseline in 2-Hour Blood Glucose Excursion During Standardized Meal Test to Week 26: Core Period
Description: 2-hour plasma glucose excursion = 2-hour PPG value minus plasma glucose value obtained 30 minutes prior to the start of meal and before investigational medicinal product (IMP) administration if IMP was injected before breakfast. Change in plasma glucose excursions were calculated by subtracting baseline value from Week 26 value. Missing data was imputed using LOCF.
Time Frame: Baseline, Week 26
Population: Analysis was performed using mITT population. Here, "overall number of participants analyzed" = participants with baseline and Week 26 assessments.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) | GLP-1 Receptor Agonist
Number analyzed (Participants) | 215 | 220
mmol/L | -1.51 (0.177) | -0.52 (0.173)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) vs GLP-1 Receptor Agonist; Analysis was performed using ANCOVA model with treatment groups, randomization strata of Week -2 HbA1c (<8.0%, >=8.0%), randomization strata of GLP-1 receptor agonist subtype (once/twice daily formulations, once weekly formulations) at screening, and world region as fixed effects and baseline 2-hour plasma glucose excursion value as a covariate. Testing according to the hierarchical testing procedure (continued only if previous endpoints were statistically significant); Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -0.99, 95% CI 2-sided [-1.468 to -0.508], Standard Error of Mean 0.244

12. Secondary Outcome: Change From Baseline in 2-Hour Blood Glucose Excursion During Standardized Meal Test to Week 52: Single Arm Extension Period
Description: 2-hour plasma glucose excursion = 2-hour PPG value minus plasma glucose value obtained 30 minutes prior to the start of meal and before IMP administration if IMP was injected before breakfast. Change in plasma glucose excursions were calculated by subtracting baseline value from Week 52 value. Missing data was imputed using LOCF.
Time Frame: Baseline, Week 52
Population: Analysis was performed on mITT population who entered the extension period. Here, "overall number of participants analyzed" = participants with baseline and Week 52 assessments.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC)
Number analyzed (Participants) | 192
mmol/L | -1.85 (0.209)

13. Secondary Outcome: Percentage of Participants Requiring Rescue Therapy During the 26 Week Treatment Period: Core Period
Description: Routine HbA1c value was used to determine the requirement of rescue medication. Threshold values at Week 12 or later on Week 12: HbA1c >8%.
Time Frame: From Baseline to Week 26
Population: Analysis was performed using mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) | GLP-1 Receptor Agonist
Number analyzed (Participants) | 252 | 253
percentage of participants | 4.8 | 15.0

14. Secondary Outcome: Percentage of Participants Requiring Rescue Therapy During the 52 Week Treatment Period: Single Arm Extension Period
Description: as for outcome 13
Time Frame: From Week 26 to Week 52
Population: Analysis was performed on mITT population who entered the extension period.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC)
Number analyzed (Participants) | 206
percentage of participants | 1.5

15. Secondary Outcome: Change From Baseline in Body Weight at Week 26: Core Period
Description: Change in body weight was calculated by subtracting baseline value from Week 26 value.
Time Frame: Baseline, Week 26
Population: Analysis was performed using mITT population. Here, "overall number of participants analyzed" = participants with baseline and at least one post-baseline body weight assessment.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) | GLP-1 Receptor Agonist
Number analyzed (Participants) | 251 | 253
kilogram (kg) | 1.89 (0.222) | -1.14 (0.220)

16. Secondary Outcome: Change From Baseline in Body Weight to Week 52: Single Arm Extension Period
Description: Change in body weight was calculated by subtracting baseline value from Week 52 value.
Time Frame: Baseline, Week 52
Population: Analysis was performed using mITT population who entered the extension period. Here, "overall number of participants analyzed" = participants with baseline and at least one post-baseline body weight assessment.
Measure: Mean (Standard Error); unit: kg
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC)
Number analyzed (Participants) | 202
kg | 2.78 (0.294)

17. Secondary Outcome: Number of Documented Symptomatic Hypoglycemia Events Per Participant-Year: Core Period
Description: Documented symptomatic hypoglycemia was an event during which symptoms of hypoglycemia were accompanied by a measured plasma glucose concentration of <=3.9 mmol/L (70 mg/dL). Hypoglycemic episodes with plasma glucose of <3.0 mmol/L (54 mg/dL) were also analyzed.
Time Frame: From Baseline to Week 26
Population: Analysis was performed on safety population which included all randomized participants who received at least one dose of open-label IMP, regardless of the amount of treatment administered. Participants were analyzed according to the treatment actually received (as treated).
Measure: Number; unit: events per participant-year
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) | GLP-1 Receptor Agonist
Number analyzed (Participants) | 255 | 256
events per participant-year
  Documented symptomatic hypoglycemia(<=3.9 mmol/L) | 1.54 | 0.08
  Documented symptomatic hypoglycemia (<3.0 mmol/L) | 0.25 | 0.01

18. Secondary Outcome: Number of Documented Symptomatic Hypoglycemia Events Per Participant-Year: Single Arm Extension Period
Description: as for outcome 17
Time Frame: From Baseline to Week 52
Population: Analysis was performed on safety population who entered the extension period and their data for whole study duration was analyzed and reported.
Measure: Number; unit: events per participant-year
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC)
Number analyzed (Participants) | 206
events per participant-year
  Documented symptomatic hypoglycemia(<=3.9 mmol/L) | 1.59
  Documented symptomatic hypoglycemia (<3.0 mmol/L) | 0.24

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of informed consent until the end of the study (up to 52 weeks).
Description: Reported AEs are treatment-emergent that is AEs that developed/worsened during during the period from the administration of first dose of the study treatments up to 3 days (9 days for the weekly GLP1) after the last administration. Analysis was performed on safety population.
Groups:
- Fixed Ratio Combination: FRC injected subcutaneously QD for 26 weeks on top of OAD therapy. Dose individually adjusted (median exposure: 183 days).
- GLP-1 Receptor Agonist: GLP-1 RA receptor agonist (liraglutide QD, exenatide BID, exenatide extended-release QW, albiglutide QW, or dulaglutide QW) injected subcutaneously for 26 weeks on top of OAD therapy. GLP-1 RAs were administered as per local labeling at the same dose schedule as prior to randomization (median exposure: 183 days).
- Fixed Ratio Combination Whole Study Period: Participants who completed core treatment period and met eligibility criteria entered in extension treatment period and received same treatment (FRC injected subcutaneously QD on top of OAD therapy) for 26 weeks (up to Week 52). Dose individually adjusted (median exposure: 365 days).
Arm/Group | Fixed Ratio Combination | GLP-1 Receptor Agonist | Fixed Ratio Combination Whole Study Period
All-Cause Mortality (participants affected / at risk) | 0/255 | 0/256 | 1/206
Serious Adverse Events (participants affected / at risk) | 10/255 | 9/256 | 21/206
Other Adverse Events (participants affected / at risk) | 69/255 | 48/256 | 75/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fixed Ratio Combination (N=255) | GLP-1 Receptor Agonist (N=256) | Fixed Ratio Combination Whole Study Period (N=206)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Duodenal Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large Intestine Polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infected Skin Ulcer (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Postoperative Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid Haemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Adenosquamous Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bladder Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Endometrial Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic Unconsciousness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Intraventricular Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Subarachnoid Haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Vasculitis Necrotising (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fixed Ratio Combination (N=255) | GLP-1 Receptor Agonist (N=256) | Fixed Ratio Combination Whole Study Period (N=206)
Diarrhoea (Gastrointestinal disorders) | 14 (14) | 6 (6) | 15 (17)
Nausea (Gastrointestinal disorders) | 22 (30) | 6 (6) | 19 (30)
Influenza (Infections and infestations) | 11 (12) | 6 (6) | 15 (19)
Nasopharyngitis (Infections and infestations) | 25 (27) | 23 (26) | 32 (37)
Upper Respiratory Tract Infection (Infections and infestations) | 9 (11) | 12 (15) | 13 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2017-05-12): https://cdn.clinicaltrials.gov/large-docs/51/NCT02787551/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-07): https://cdn.clinicaltrials.gov/large-docs/51/NCT02787551/SAP_001.pdf